CLINICAL TRIAL: NCT05978583
Title: Assessing the Impact of Physical and Occupational Therapy for Patients Admitted for Bone Marrow Transplant on Outcomes
Brief Title: Impact of Physical and Occupational Therapy in New BMT Patients
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2252
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Bone Marrow Transplantation; Bone Marrow Disease
Keywords: exercise; physical therapy
MeSH Terms: conditions — Bone Marrow Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- physical and occupational therapy: Physical and occupational therapy consultation might be used to provide targeted prehabilitation interventions.

SUMMARY:
This is a single-site, non-randomized, observational study designed to evaluate the impact of adding physical and occupational therapy consultation upon inpatient admission for a bone marrow transplantation (BMT). The purpose of this study is to investigate whether consultation with physical and occupational therapists as part of the general admission order set for patients scheduled for bone marrow transplant will result in reduced complications, morbidity, length of inpatient stay, 30-day readmission, and 90-day mortality. Baseline data collection will be used to determine eligibility. This study will be partially retrospective (pre-implementation of physical and occupational therapy consultation order) and partially prospective.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of admission for bone marrow transplantation (BMT)
2. Received BMT

Exclusion Criteria:

1. No history of inpatient admission for BMT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are admitted for bone marrow transplantation (BMT) at the study site.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
30-day readmission | Up to 30 days after bone marrow transplantation
  30-day readmission rates will be calculated using historical data (pre-intervention) and compared to rates once physical and occupational therapy consultation has been included in the inpatient admission order set for bone marrow transplantation (BMT).

SECONDARY OUTCOMES:
The feasibility | 1 day (the date of bone marrow transplantation)
  The proportion of individuals who received a physical and occupational therapy consultation in the prospective group.
Acute care length of stay | Up to 90 days after bone marrow transplantation
  Acute care length of stay will be calculated using historical data (pre-intervention) and compared to rates once physical and occupational therapy consultation has been included in the inpatient admission order set for BMT.
Mortality rates | Up to 90 days after bone marrow transplantation
  Mortality rates will be calculated by comparing, how many subjects died pre-intervention and post-intervention, using medical record data.
Complication types and rates | Up to 90 days after bone marrow transplantation
  Complication types and rates will be calculated and compared pre-intervention and post-intervention using medical record data.

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Stephen, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comphrehensive Cancer Center at University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials